CLINICAL TRIAL: NCT03714425
Title: Efficacy of the Quell Wearable Device for Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Robert N. Jamison, PhD, Professor of Anaesthesia, Harvard Medical School, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018P002392
Record Dates: First submitted 2018-10-17; First posted 2018-10-22 (Actual); Results first posted 2022-06-21 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-07

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Intervention Model Description: High frequency device vs. Low frequency device
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- High frequency device (Active Comparator): Subjects will use high frequency Quell devices.
  Interventions: Device: Quell
- Low frequency device (Sham Comparator): Subjects will use low frequency Quell devices.
  Interventions: Device: Quell

INTERVENTIONS:
Device: Quell — Quell is a Transcutaneous Electrical Nerve Stimulator Device (TENS). The device will use nerve stimulation to treat chronic pain by sending signals to the brain that cause it to release natural opioids.

SUMMARY:
This study is designed for patients with primary fibromyalgia (FM) pain. The overall aim of the study is to determine the effect of the high frequency Quell device to manage FM compared with a low frequency device. Investigators hypothesize that those assigned to using the high frequency Quell device will report reduced pain compared with those using the low frequency Quell device; with those using the high frequency device also showing more improvement in sleep, mood, and level of activity. Investigators also hypothesize that frequency of using the Quell (increased tolerability and adherence) will be correlated with greater reduction in pain.

DETAILED DESCRIPTION:
The Quell is battery powered with rechargeable batteries and is strapped to participant's upper calf with a velcro band. It has been cleared by the FDA for safety. It is designed to improve fibromyalgia by the principles of transcutaneous electrical stimulation of nerves much like a traditional transcutaneous electrical nerve stimulator (TENS) unit. Investigators expect to enroll approximately 130 subjects in this study. Participants will be equally randomized to one of two experimental groups: High Frequency Quell group (N=65) or Low Frequency Quell group (N=65). This study hopes to find out whether low frequency or high frequency stimulation is most useful among persons with fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

1. have chronic pain related to FM for > 3 months' duration
2. average 4 or greater on a pain intensity scale of 0 to 10
3. are able to speak and understand English
4. have a smartphone (Android or iPhone)

Exclusion Criteria:

1. diagnosis of cancer or any other malignant disease
2. acute osteomyelitis or acute bone disease
3. present or past DSM-V diagnosis of schizophrenia, delusional disorder, psychotic disorder, or dissociative disorder that would be judged to interfere with study participation
4. pregnancy
5. any clinically unstable systemic illness judged to interfere with treatment
6. a pain condition requiring urgent surgery
7. an active substance use disorder, such as cocaine or IV heroin use (positive on the Mini International Neuropsychiatric Interview; M.I.N.I. v.5.0), that would interfere with study participation
8. have an implanted cardiac pacemaker, defibrillator, or other implanted device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Chestnut Hill, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jamison RN, Edwards RR, Curran S, Wan L, Ross EL, Gilligan CJ, Gozani SN. Effects of Wearable Transcutaneous Electrical Nerve Stimulation on Fibromyalgia: A Randomized Controlled Trial. J Pain Res. 2021 Jul 24;14:2265-2282. doi: 10.2147/JPR.S316371. eCollection 2021. PMID 34335055

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | High Frequency Device | Low Frequency Device
Started | 62 | 57
Completed | 55 | 46
Not Completed | 7 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Frequency Device | Low Frequency Device | Total
Number analyzed (Participants) | 62 | 57 | 119
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 57 | 52 | 109
  >=65 years | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.3 (13.1) | 52.3 (13.8) | 50.4 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 53 | 111
  Male | 4 | 4 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 5 | 10
  White | 48 | 47 | 95
  More than one race | 7 | 4 | 11
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 62 | 57 | 119

OUTCOME MEASURES:

1. Primary Outcome: Patients' Global Impression of Change
Description: The questionnaire reflects a patient's belief about the efficacy of treatment. The Patients' Global Impression of Change (PGIC) is a 7-point scale (1-7) depicting a patient's rating of overall improvement. Patients rate their change as 1="very much improved," 2="much improved," 3="minimally improved," 4="no change," 5="minimally worse," 6="much worse," or 7="very much worse." Lower values represent a better outcome.
Time Frame: 3 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | High Frequency Device | Low Frequency Device
Number analyzed (Participants) | 62 | 57
score on a scale | 3.58 [3.09 to 4.07] | 3.24 [2.74 to 3.75]

2. Secondary Outcome: The Brief Pain Inventory
Description: The Brief Pain Inventory assesses the severity of pain and its impact on functioning. Pain Severity Score is calculated by adding the scores for questions 2, 3, 4 and 5 and then dividing by 4. This gives a severity score out of 10 (0-10), where 0 means no pain and 10 is worst possible pain. Pain Interference Score is calculated by adding the scores for questions 8a, b, c, d, e, f and g and then dividing by 7. This gives an interference score out of 10 (0-10), where 0 means does not interfere and 10 means completely interferes. Lower values represent a better outcome.
Time Frame: Baseline, 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Frequency Device | Low Frequency Device
Number analyzed (Participants) | 62 | 57
score on a scale | 5.8 (1.6) | 5.5 (1.5)

3. Secondary Outcome: Revised Fibromyalgia Impact Questionnaire
Description: The Revised Fibromyalgia Impact Questionnaire (FIQR) is an assessment and evaluation instrument developed to measure fibromyalgia (FM) patient status, progress and outcomes. The FIQR has 3 domains: function, overall impact and symptoms. FIQR has 21 individual questions and all questions are based on an 11-point numeric rating scale of 0 to 10, with 10 being 'worst'. The summed score for function (range 0 to 90) is divided by 3, the summed score for overall impact (range 0 to 20) is not changed, and the summed score for symptoms (range 0 to 100) is divided by 2. The total FIQR is the sum of the three domain scores. The total score of the FIQR ranges from 0 to 100. Lower values represent a better outcome.
Time Frame: Baseline, 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Frequency Device | Low Frequency Device
Number analyzed (Participants) | 62 | 57
score on a scale | 61.3 (16.3) | 52.8 (17.3)

4. Secondary Outcome: Pain Catastrophizing Scale
Description: The Pain Catastrophizing Scale (PCS) instructions ask participants to reflect on past painful experiences, and to indicate the degree to which they experienced each of 13 thoughts or feelings when experiencing pain, on 5-point scales with the end points (0) not at all and (4) all the time. The total score is computed by summing responses to all 13 items (scale 0-4). PCS total scores range from 0 - 52. The higher the score, the more catastrophizing thoughts are present. Lower values represent a better outcome.
Time Frame: Baseline, 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Frequency Device | Low Frequency Device
Number analyzed (Participants) | 62 | 57
score on a scale | 21.5 (13.2) | 17.8 (12.3)

5. Secondary Outcome: Pain Disability Index
Description: The Pain Disability Index is a simple and rapid instrument for measuring the impact that pain has on the ability of a person to participate in essential life activities. The total score is a sum of all 7 categories of life activity listed. A score of 0 means no disability at all, and a score of 10 signifies that all of the activities in which people would normally be involved have been totally disrupted or prevented by the pain. The total index ranges from 0 to 70. The higher the index the greater the person's disability due to pain. Lower values represent a better outcome.
Time Frame: Baseline, 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Frequency Device | Low Frequency Device
Number analyzed (Participants) | 62 | 57
score on a scale | 39.4 (15.6) | 34.6 (15.5)

6. Secondary Outcome: Hospital Anxiety and Depression Scale
Description: The Hospital Anxiety and Depression Scale (HADS) was developed to assess depression and anxiety in patients. Responses are rated on a scale from 0 to 3, with higher scores indicating higher severity. The ratings of the 14 items are summed to yield a total score (0 to 42), or for each subscale separately (0 to 21). 0 to 7 for normal or no anxiety/depression, 8 to 10 for mild, 11 to 14 for moderate, and 12 to 21 for severe anxiety/depression. Lower values represent a better outcome.
Time Frame: Baseline, 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Frequency Device | Low Frequency Device
Number analyzed (Participants) | 62 | 57
score on a scale | 18.5 (7.3) | 15.8 (7.6)
Statistical Analysis 1: Comparison: High Frequency Device vs Low Frequency Device; Test type: Superiority; p < 0.05, t-test, 2 sided — The primary research objective to measure perceived improvement in pain at three months was assessed using a two-sample t-test of PGIC scores between the two treatment groups using a type I error rate of 0.05 (two-sided); Most of the analyses involved delta scores reflecting changes within subjects, though we compared PGIC raw scores rather than change scores

7. Secondary Outcome: Helpfulness Rating
Description: Self-report rating "How helpful was the TENS for your fibromyalgia?" 0=not at all helpful, 10=very helpful.
Time Frame: Post-treatment at 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Frequency Device | Low Frequency Device
Number analyzed (Participants) | 62 | 57
score on a scale | 4.8 (3.5) | 4.8 (2.6)

ADVERSE EVENTS:
Time Frame: 3 months
Description: Adverse events list
Groups:
- High Frequency Device: High frequency active device
- Low Frequency Device: Low frequency sham device
Arm/Group | High Frequency Device | Low Frequency Device
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/57
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/57
Other Adverse Events (participants affected / at risk) | 0/62 | 0/57

LIMITATIONS AND CAVEATS:
There were several limitations. The study included a limited number of subjects. Subjects were only followed for 3 months. There was no in-person history or physical examination. Many chose not to tolerate the higher levels of stimulation. The subjects had other medical comorbidities. The symptom reporting was not required while the participants were using the TENS.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-27): https://cdn.clinicaltrials.gov/large-docs/25/NCT03714425/Prot_SAP_001.pdf